CLINICAL TRIAL: NCT03133052
Title: The CTA-MCI Study: a Randomized Controlled Clinical Trial to Evaluate the Effect of Cognitive Control Training on Episodic Memory Function in Patients With Amnestic Mild Cognitive Impairment
Brief Title: CTA-MCI: Cognitive Control Training in Patients With Amnestic Mild Cognitive Impairment(CTA-MCI)
Acronym: CTA-MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTCI-cognitive training
Record Dates: First submitted 2017-04-01; First posted 2017-04-28 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Amnestic Mild Cognitive Impairment
Keywords: cognitive control training; aMCI; MRI; RCT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Active Comparator): Intervention: Internet-based adaptive cognitive control training program. 5 x 30 minutes per week, for 12 weeks.
  Interventions: Behavioral: internet-based adaptive cognitive control training program
- control group (Placebo Comparator): Intervention: placebo program: a fixed, primary difficulty level task. 5 x 30 minutes per week, for 12 weeks.
  Interventions: Behavioral: placebo program

INTERVENTIONS:
Behavioral: internet-based adaptive cognitive control training program — The cognitive training will be an internet-based adaptive cognitive control training program, specific training paradigms include Flanker, 1-back, 2-back. To maintain task difficulty, the tasks will be grouped based on the task difficulty. Furthermore, each task will have various difficulty levels.
  Arms: training group
Behavioral: placebo program — For the control group, a fixed, primary difficulty level program for all participants is set.
  Arms: control group

SUMMARY:
This study evaluates the efficacy and mechanism of internet-based cognitive control training on episodic memory function in patients with amnestic Mild Cognitive Impairment(aMCI). Half of participants will receive adaptive internet-based cognitive control training program, while the other half will receive a fixed, primary difficulty level task.

DETAILED DESCRIPTION:
Background:

Alzheimer's disease (AD) is a common dementia in elderly populations, and amnestic mild cognitive impairment (aMCI) refers to a transitional stage between normal aging and early dementia. Patients with aMCI are at higher risks of evolving toward AD. Although it has been widely recognized that early intervention of aMCI holds the potential to delay or even reverse the cognitive impairment, no treatment is available yet. Episodic memory dysfunction is the characteristic impairment in aMCI, cognitive control training significantly improved executive function in patients with aMCI . Whether and how cognitive control training improves episodic memory function in patients with aMCI remains largely unknown.

Objectives:

The primary objective of this double-blinded, randomized RCT is to assess whether internet-based cognitive control training in patients with amnestic Mild Cognitive Impairment improves their episodic memory function. The second objective is to evaluate the effect of cognitive control training on neural plasticity, including brain activation and white matter integrity, which are assessed by functional and structural MRI.

Patients and Methods:

The proposed study is a single-center, double-blinded, randomized controlled trial that will include 70 patients diagnosed with aMCI from the neurology clinics at The First Affiliated Hospital, Zhejiang University. The patients will be randomized to either a training or a control group. The intervention is internet-based cognitive control training performed for 30 minutes over 60 sessions. Neuropsychological assessment and functional magnetic resonance imaging (MRI) will be performed before and 12 weeks after training.

Relevance:

Currently there is no known treatment available for aMCI. The proposed study is to determine the efficacy of cognitive control training on episodic memory function in patients with aMCI. Secondly, using functional and structural MRI, this study is to reveal the potential mechanism underlying cognitive control training.

ELIGIBILITY:
Inclusion Criteria:

* Literate Chinese, aged 50 years and older
* Complaint about memory loss and confirmed by an informant
* Cognitive impairment in memory domain, adjusted for age and education
* Normal or near-normal performance on general cognitive function and no or minimum impairment of daily life activities
* Clinical dementia rating (CDR) =0.5, Mini-Mental State Examination (MMSE) score ≥ 20 (primary school) or ≥ 24 (junior school or above)
* Failure to meet the criteria for dementia

Exclusion Criteria:

* history of clinically significant stroke
* neurological diseases that may lead to neurological distortion, including schizophrenia, severe anxiety or depression, frontotemporal dementia，Huntington disease, brain tumor, parking disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal pressure hydrocephalus
* systemic diseases that may lead to neurological distortion, including hypothyroidism, folic acid deficiency, vitamin B12 deficiency, severe anemia, specific infection such as HIV and syphilis
* clinically significant gastrointestinal, renal, hepatic, respiratory, endocrine, or cardiovascular system disease;
* cancer, alcoholism, drug addiction;
* severe aphasia, physical disabilities, or any other factor that may preclude completion of neuropsychological testing;
* use of medications that may affect cognitive functioning, including tranquilizers, anti-anxiolytics, hypnotics, nootropics, and cholinomimetic agents;
* inability to undergo a brain MRI.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-07-09 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 12 weeks
  The study uses MoCA to assess changes in the global cognitive function after an intervention of cognitive control training
Auditory Verbal Learning Test (AVLT) | 12 weeks
  The study uses AVLT to assess changes in the episodic memory function after an intervention of cognitive control training

SECONDARY OUTCOMES:
Gray matter volume | 12 weeks
  The study uses voxel-based morphometry (VBM) to measure changes of gray matter volume after an intervention of cognitive training.
White matter Integrity | 12 weeks
  The study uses Diffusion tensor imaging and tracking (DTI) to measure changes of the Integrity of white matter after an intervention of cognitive control training
Brain response change | 12 weeks
  The study uses task functional MRI (fMRI) to measure the brain response changes during the task after an intervention of cognitive control training
Functional connectivity across regions | 12 weeks
  The study uses resting state functional MRI(rs-fMRI) and task fMRI to measure changes of functional connectivity across regions after an intervention of cognitive control training

OTHER OUTCOMES:
MoCA | 6 months
  The participants will be followed up 6 months after recruitment. The training is not mandatory after 12 weeks, but the training details will be acquired from the online system.
AVLT | 6 months
  The participants will be followed up 6 months after recruitment. The training is not mandatory after 12 weeks, but the training details will be acquired from the online system.
Gray matter volume | 6 months
  The participants will be followed up 6 months after recruitment. The training is not mandatory after 12 weeks, but the training details will be acquired from the online system.
White matter Integrity | 6 months
  The participants will be followed up 6 months after recruitment. The training is not mandatory after 12 weeks, but the training details will be acquired from the online system.
Functional connectivity across regions | 6 months
  The participants will be followed up 6 months after recruitment. The training is not mandatory after 12 weeks, but the training details will be acquired from the online system.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Ph.D., Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang K, Wang J, Peng G, Liu P, He F, Zhu Z, Luo B. Effect of cognitive training on episodic memory retrieval in amnestic mild cognitive impairment patients: study protocol for a clinical randomized controlled trial. Trials. 2019 Jan 8;20(1):26. doi: 10.1186/s13063-018-3143-0. PMID 30621794